CLINICAL TRIAL: NCT04399083
Title: Real-Time Caffeine Optimization During Total Sleep Deprivation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Principal Investigator, William D. Killgore, Professor, University of Arizona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1912215022
Record Dates: First submitted 2020-02-04; First posted 2020-05-22 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Caffeine; Sleep Deprivation; Shift-Work Related Sleep Disturbance
MeSH Terms: conditions — Sleep Deprivation | interventions — Caffeine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Dietary Supplement: Caffeine

INTERVENTIONS:
Dietary Supplement: Caffeine — Caffeine will be administered to each participant following an individualized optimal dosing schedule created by the 2B-Alert app. Individualized caffeine dosing schedules will be created by the 2BAlert app on the smartphone the participant uses to do Smart-PVT tests. Study staff will run the optimization at 1900 on Day 15. The algorithm will recommend caffeine dosing to optimize performance during the Peak Alertness window (e.g. from 0300-0900 on Day 16, 44-50 hours of continuous sleep loss). Doses could be recommended at any hour from 2000 on Day 15 to 0800 on Day 16. HOWEVER, the algorithm will not exceed 800 mg of caffeine across the entire study AND it will not dose more than 300 mg of caffeine at a time. Gum will be chewed for a total of 10 minutes by each participant and then discarded.
  As there will be no placebo in this protocol, randomization and blinding procedures are not necessary. IT IS IMPORTANT TO NOTE THAT SOME PARTICIPANTS MAY NOT RECEIVE CAFFEINE AT ALL.

SUMMARY:
Sleep deprivation (SD) has a powerful degrading effect on cognitive performance, particularly psychomotor vigilance (PV) and reaction time. Caffeine is well known to be an effective countermeasure to the effects of SD. However, individuals differ in both their response to SD and to the administration of caffeine. This has made it difficult to provide individualized recommendations regarding the use of caffeine to sustain alertness when needed. For the past two decades, the Army's Biotechnology HPC Institute (BHSAI), in collaboration with the Walter Reed Army Institute of Research, have been developing statistical models to predict individual performance during prolonged SD. Recently, this resulted in the publication of the 2B-Alert app, a computer algorithm based on large datasets that can learn an individual's response to SD by combining actigraphic sleep data with simultaneously acquired PV performance data. The 2B-Alert algorithm can predict an individual's sleep need and performance after ~2 weeks of training the model. Recently, the model has been extended to incorporate individualized responses to caffeine. This was recently validated in a retrospective study published by BHSAI in 2019. The present study is designed to test the predictive capacity of the 2B-Alert app in real time. During Phase 1 a total of 21 healthy participants will wear an actigraph & complete multiple daily PV tests on a personal cell phone. After 2 weeks, these individuals will attend Phase 2 involving an in-laboratory stay & SD. Participants will have an 8-hour period of sleep in the laboratory, followed by 62 hours of continuous wakefulness. During these 62 hours, participants will complete PV and mood testing every 3 hours. The 2B-Alert app will be used to predict individual caffeine need to sustain performance at near-baseline levels based on the statistical model. At 44 hours SD, participants will undergo a 6-hour "alertness window" where they may receive individualized doses of caffeine based on the recommendations of the model. After 62 hours of SD, Phase 3 begins, involving a night of monitored recovery sleep and additional sessions of PV and mood testing until release from the study at 6 pm on the final day. It is hypothesized that the 2B-Alert app will be effective at providing caffeine dosing recommendations that return PV and mood performance to normal levels during the alertness window.

DETAILED DESCRIPTION:
The first objective of the present study is to determine whether the 2B-Alert Caffeine Optimization Model (2BAlert) can create individualized caffeine schedules that effectively recover PVT performance during a specified window of time. The 2BAlert model is the linchpin of the comprehensive fatigue management system being developed by Walter Reed Army Institute of Research (WRAIR) and Biotechnology High Performance Computing Software Applications Institute (BHSAI). It is a software tool that "learns" (quantifies) the relationship between an individual's sleep/wake parameters (as objectively measured via wrist actigraphy) and his/her psychomotor performance (as objectively measured on a PVT). It quantifies the extent to which an individual is sensitive/resilient to the effects of sleep loss, and produces individualized performance predictions that can be used to inform decisions regarding current and future readiness, as well as the application of fatigue countermeasures such as naps or caffeine. The most recent version of 2BAlert can apply fatigue countermeasures directly to an individual based on their individualized performance prediction. This model gives recommendations for when and how much caffeine to use in order to optimize performance during a specified period of time. While this model has been applied post-hoc to previously collected data, it has yet to be tested in real-time. This study will provide the first opportunity to directly test if the model can be effectively used, in real-time, to recover PVT performance to a desired level (i.e., 275ms) when required (i.e., a six hour period following 44 hours of sleep loss).

A second objective of the present study is to investigate if 2BAlert can not only recover PVT performance during a specified period, but also recover increases in self-reported stress and anxiety related to sleep-loss. Data from a previous study by WRAIR shows that self-reported stress and anxiety increase after 1 night of sleep loss and continues to increase after a second night of continuous sleep deprivation. These measures return to baseline following 12 hours of recovery sleep and map directly onto PVT performance. Therefore, the investigators hypothesize that if PVT performance can be recovered by caffeine, self-reported stress and anxiety can also return close to baseline levels with caffeine.

A tertiary objective of the study is to assess whether images acquired using a smartphone camera are suitable for developing a passive, non-intrusive computer-vision system that could substitute the PVT for assessing alertness. Currently, the algorithm uses PVT data because: (a) compared to other performance measures, the PVT is relatively sensitive to sleep loss and the circadian rhythm of alertness; and (b) there are no learning effects on the PVT. However, the PVT requires an individual to actively engage in a 3- to 10-min long test, which must be performed at least a dozen times during sleep deprivation, making it a sensitive but impractical test to measure a Soldier's alertness in operational settings.

All participants will participate in the following continuous study phases. Caffeine gum may be administered during this study.

Phase 1: At Home Sleep/Wake Measurement: All participants will be instructed to maintain their normal sleep/wake schedule for the 13 days/12 nights immediately preceding phase 2 (the in-laboratory portion of the study). Compliance will be verified objectively via wrist actigraphy. Participants will be given a smartphone and asked to complete a PVT on it every 3 hours while awake and log their normal caffeine use as well as daily sleep duration.

Phase 2: In-Laboratory Sleep/Wake and PVT Performance Assessment: Participants will report to the sleep lab at 1900 hrs on Day 13. While awake in the laboratory, they will complete various cognitive tests, including the PVT, and record a 3-minute video of their face every 3 hours. They will be allowed to sleep from 2300 hrs on Day 13 until 0700 hrs on Day 14 and sleep will be monitored via PSG and actigraphy. This will be followed by 62 hours of continuous wakefulness (i.e., from 0700 hrs on Day 14 until 2100 hrs on Day 16). At 1900 on Day 15, 2BAlert will be run for each individual and will use each individual's previous sleep and performance to create an individualized caffeine dosing schedule to optimize performance from 0300-0900 on Day 16.

Phase 3: In-Laboratory Recovery: All participants will undergo a recovery phase consisting of 12 hours time in bed from 2100 hrs on Day 16 until 0900 hrs on Day 17 & sleep will be monitored via PSG and actigraphy. The cognitive testing and facial video recording schedule will continue from Phase 2 during wake hours. After being evaluated by a study physician they will be released from the study at approximately 1800 hrs on Day 17. Thus, participants will be in the laboratory for a total of 95 hours.

The main endpoint for this study is psychomotor vigilance test performance (PVT), measured using Smart-PVT. A secondary endpoint is self-reported stress and anxiety, as measured by the Stress Visual Analog Scale and the Spielberger State-Trait Anxiety Inventory, respectively. A third endpoint of the study is to test if facial images captured with the phone camera could be used to assess the alertness level of subjects under sleep deprivation.

Hypotheses to be tested: (a) Psychomotor performance data collected on the Smart-PVT will stay at or below 275ms during the Peak Alertness Window of optimized performance thus indicating that 2BAlert is valid and ready to be utilized in future field studies and operational settings. (b) Self-reported stress and anxiety will return to baseline levels during the Peak Alertness Window and map onto the recovery of PVT performance during this time window.

BACKGROUND: Sleep loss-induced neurobehavioral deficits are a recognized threat to safety and productivity in both civilian and military operational settings. Highly-publicized fatigue-related accidents and mishaps (including commercial mishaps such as those occurring at 3-Mile Island, Chernobyl, and Bhopal; and military mishaps such as the ambush of the 507th Maintenance Company) continue to draw attention to the problem of sleep loss/sleepiness in operational environments. Such accidents highlight detrimental effects of sleep loss on decision-making, vigilance, problem-solving and other mental abilities critical to military effectiveness. Publications and manuals from the Army, U.S. Marine Corps, and the U.S. Navy have documented militarily-relevant deleterious effects of sleep loss on alertness and performance. The Army's fifth Mental Health Advisory Team survey of Warfighters serving in Operation Iraqi Freedom and Operation Enduring Freedom revealed that service members who reported less sleep also reported higher rates of accidents and mistakes, and more frequently endorsed negative mental health items.

The Department of Defense has funded development of a computational model for quantifying the effects of daily sleep amounts on neurobehavioral performance. The most recent (and most advanced) version of the mathematical sleep/performance prediction model is the 2BAlert model, developed by BHSAI. Like its predecessors, 2BAlert was based primarily on PVT data collected in the WRAIR sleep research laboratory. PVT data was used because, for the purpose of constructing sleep/performance prediction models, it is generally superior to data from other performance measures in several important respects: (a) compared to other performance measures, the PVT is relatively sensitive to sleep loss and the circadian rhythm of alertness; (b) there are no learning effects on the PVT; and (c) it has previously been demonstrated that a PVT-based sleep/performance prediction model has good ecological validity. That is, the PVT-based model predictions of performance effectiveness have been shown to correlate well with 'risk of accidents' in actual railroad operations.

The current 2BAlert tool comes in two forms: 1)a web-based tool that takes sleep and caffeine schedules and displays the predicted GROUP AVERAGE performance & 2)a smartphone app that utilizes individual performance measured with the PVT on a smartphone to individualize the performance predictive model. This version of the tool was successfully validated in a recent study by WRAIR. The most recent version of the smartphone app uses individualized performance predictions to compute individualized caffeine scheduling that optimize performance during specific periods. While this tool was developed using data collected at WRAIR and has been run post-hoc on data previously collected at WRAIR, it has yet to be tested in real-time. Therefore, the purpose of this study is to validate this caffeine optimization algorithm in real-time. The investigators will be utilizing the same study protocol as the recent WRAIR study because it is known there is variability in performance in a healthy population over this time period and that overall performance is slower than 275ms and self-reported stress and anxiety increase significantly without a caffeine intervention. Additionally, by utilizing a previous study design the investigators can minimize the burden on the study team in creating new documentation and schedules.

Taking a step back, it is important to address why caffeine optimization is important and relevant for the military. While caffeine is widely accepted and utilized as a stimulant to counter the effects of fatigue associated with shift work and sleep loss, a previous study conducted by WRAIR has shown that caffeine loses its effectiveness and can even slow recovery with repeated use and chronic sleep loss. This surprising result indicates that caffeine has a limit and a cost, and, therefore, the Warfighter would be more effective if he or she utilized caffeine optimally. For previous caffeine studies with similar lengths of continuous sleep deprivation as the current protocol, participants were given 800mg of caffeine during each night. While this research suggests that the investigators could recover performance by giving all participants in this study 800mg of caffeine, the 2BAlert algorithm will allow the investigators to give some participants less caffeine but still reach the same outcome as if everyone had been given 800mg of caffeine.

Recent research applied the 2BAlert algorithm post-hoc using parameters laid out in this protocol. The model results show that all participants recovered performance during the Peak Alertness Window, i.e. between 44-50 hours awake, where recovery is defined as 275ms or faster, and over half the subjects required less than half the max total allowable amount of caffeine (800mg), while three subjects required no caffeine at all. The investigators hope to validate 2BAlert by applying it to real-time data utilizing the original study design.

In addition to testing the Caffeine Optimization model, the investigators are also interested in testing the hypothesis that if PVT performance can be recovered with caffeine, self-reported stress and anxiety can also be recovered. Recent work found that self-reported stress and anxiety increased with increased sleep loss and recovered to baseline after recovery sleep, following the same trend as PVT performance data. While previous work has shown that self-reported stress and anxiety increase with 1 night of sleep loss, these are the first data to show that self-reported stress and anxiety continue to increase after 2 nights of sleep loss. There are currently no studies reporting if and how self-reported stress and anxiety can be recovered with caffeine during sleep loss.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and non-pregnant, non-lactating women.
* Must demonstrate adequate comprehension of the protocol by achieving a score of at least 80% correct on a short multiple-choice quiz. Individuals who fail to achieve a passing score on the initial quiz will be given one opportunity to retest after a review of protocol information. Individuals who fail the comprehension assessment for the second time will be disqualified

Exclusion Criteria:

* Self-reported habitual nightly sleep amounts outside the target range of approximately 6-9 hours (i.e., less than 6 hours per night or more than 9 hours per night, on average)
* Self-reported nighttime lights-out times earlier than approximately 2100 hours on average during weeknights (Sunday through Thursday)
* Self-reported morning wake-up times later than approximately 0900 on average during weekdays (Monday through Friday)
* Self-reported habitual napping (> 3 times per week) in conjunction with normal sleep habits
* Self-reported symptoms suggestive of a sleep disorder (to include but not limited to sleep disordered breathing/sleep apnea, narcolepsy, idiopathic hypersomnia, restless leg syndrome, parasomnias, REM behavior disorder, etc.)
* History of a sleep disorder (to include all of the above)
* Any use of prescription or over-the-counter sleep aids during the 6 month period prior to screening indicative of a potential sleep disorder as determined by the examining study physician (e.g., use of a sleep aid for several nights following time zone travel, or the occasional use of a sleep inducing medication (e.g. 1-2 times per month), would not necessarily constitute evidence of a sleep disorder and result in disqualification)
* Self-reported caffeine use in excess of 400 mg (e.g., approximately 8 caffeinated sodas or approximately 3-4 12-oz cups of coffee) per day on average
* History of neurologic disorder (to include but not limited to epilepsy or another seizure disorder, amnesia for any reason, hydrocephalus, MS). An infrequent or resolved single neurological event (e.g., childhood seizure, rare sporadic migraine headaches, resolved meningeal infection with no sequelae) may be deemed non-exclusionary at the discretion of the examining study physician.
* Score of 14 or above on the Beck Depression Inventory
* Score of 41 or above on the Spielberger Trait Anxiety Inventory
* Score of lower than 31 or higher than 69 on the Morningness-Eveningness Questionnaire
* Self-reported or suspected regular nicotine use (or addiction) (defined as more than 1 cigarette or equivalent per week) within the last 1 year)
* Self-reported or suspected heavy alcohol use (minimum limit to define heavy alcohol use is 14 drinks per week or as determined by the examining study physician)
* History of cardiovascular disease (to include but not limited to arrhythmias, valvular heart disease, congestive heart failure, history of sudden cardiac death or myocardial infarction)
* Underlying acute or chronic pulmonary disease requiring daily inhaler use
* Kidney disease or kidney abnormalities
* Liver disease or liver abnormalities
* Self-reported history of psychiatric disorder requiring hospitalization or use of psychiatric product for any length of time
* Self-reported or suspected use of products or drugs that cannot be safely discontinued during in-laboratory phases, to be determined on a case-by-case basis by the examining study physician
* Self-reported or suspected current use of other illicit drugs (to include but not limited to benzodiazepines, amphetamines, cocaine, marijuana)
* (Females only) Positive urine pregnancy result
* (Females only) Self-reported or suspected current breast-feeding or collecting breast-milk
* Resting blood pressure above 140/90 or resting pulse > 110 beats per minute Note that if a repeat measurement is within range, volunteer will not be excluded.
* BMI ≥ 30 (Obese Class I or greater)
* Clinically significant values (as determined by the reviewing study physician) for any hematology or chemistry parameter. Reviewing study physician may opt to repeat any clinically significant tests and include participants whose repeat test values are not clinically significant.
* Positive urine nicotine/cotinine result during screening visit
* Positive urine drug result during screening visit
* Positive saliva alcohol results during screening visit
* Inability to read and sign consent
* Failure to obtain required approved official leave to participate.
* Failure to cooperate with requirements of the study, e.g. failure to complete 80% of Smart-PVTs during Phase 1 (Days 2-13)

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Changes in Psychomotor Vigilance Tests (PVT) Reaction Time During Peak Alertness Window following 44 hours of continuous wake | Task duration is 5 minutes. Task will occur hourly from 2130 on Day 15 to 0930 on Day 16.
  Assesses the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness Subjects continuously monitor a blank display and touch the smart phone screen as quickly as possible in response to a visual stimulus (i.e. a millisecond counter that begins at zero and stops when you press the button). Outcome measures: Mean RT (ms), Mean Speed (s-1), Lapses (#) The primary objective of this study is to determine if the real-time 2B-Alert Caffeine Optimization algorithm can produce personalized recommendations that will keep individual performance at or below 275 ms (milliseconds) for all study participants throughout a 6-hour Peak Alertness Window following 44 hours of continuous wake
Changes in Psychomotor Vigilance Tests (PVT) Reaction Time Phase 1 at home monitoring | Task duration is 5 minutes. Every 3 hours during Phase 1 (Days 2 - 13: at 0800, 1100, 1400, 1700, 2000, and 2300 hrs)
  Assesses the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness Subjects continuously monitor a blank display and touch the smart phone screen as quickly as possible in response to a visual stimulus (i.e. a millisecond counter that begins at zero and stops when you press the button). Outcome measures: Mean RT (ms), Mean Speed (s-1), Lapses (#)
Changes in Psychomotor Vigilance Tests (PVT) Reaction Time Phase 2 sleep deprivation not including Peak Alertness Window | Task duration is 5 minutes. Every 3 hours Phase 2 Day 14 at 0930, 1230, 1530, 1830, 2130; Day 15 at 0000, 0330, 0630, 0930, 1230, 1530, 1830; Day 16 at 1230, 1530, 1830
  Assesses the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness Subjects continuously monitor a blank display and touch the smart phone screen as quickly as possible in response to a visual stimulus (i.e. a millisecond counter that begins at zero and stops when you press the button). Outcome measures: Mean RT (ms), Mean Speed (s-1), Lapses (#)
Changes in Psychomotor Vigilance Tests (PVT) Reaction Time Phase 3 recovery | Task duration is 5 minutes. Every 3 hours Phase 3 Day 17 at 0930, 1230 and 1530.
  Assesses the effects of sleep loss on visual reaction time as a behavioral measure of sleepiness Subjects continuously monitor a blank display and touch the smart phone screen as quickly as possible in response to a visual stimulus (i.e. a millisecond counter that begins at zero and stops when you press the button). Outcome measures: Mean RT (ms), Mean Speed (s-1), Lapses (#)

SECONDARY OUTCOMES:
Stress Visual Analog Scale Phase 2 Sleep Deprivation | Task duration ~15 seconds. Every 3 hours starting Day 14 at 0930 until Day 16 1830.
  Measures stress on a sliding scale from not stressed to very stressed. Choose the level of stress that most closely corresponds to your current level of stress by using the mouse to slide the marker between not stressed and very stressed. Outcome measure: stress level (0-100).
Stress Visual Analog Scale Phase 3 Recovery | Task duration ~15 seconds. Every 3 hours on Day 17 at 0930, 1230, and 1530.
  Measures stress on a sliding scale from not stressed to very stressed. Choose the level of stress that most closely corresponds to your current level of stress by using the mouse to slide the marker between not stressed and very stressed. Outcome measure: stress level (0-100).
Spielberger State-Trait Anxiety Inventory - State (STAI-S) Phase 2 Sleep Deprivation | Task duration ~3 minutes. Every 3 hours starting Day 14 at 0930 until Day 16 1830.
  Used to identify state changes in anxiety in healthy adults. Volunteers are instructed to rate on a 4-point scale how closely they identify with 20 statements related to state anxiety. Outcome measure: state anxiety level (20-80).
Spielberger State-Trait Anxiety Inventory - State (STAI-S) Phase 3 Recovery | Task duration ~3 minutes. Every 3 hours on Day 17 at 0930, 1230, and 1530.
  Used to identify state changes in anxiety in healthy adults. Volunteers are instructed to rate on a 4-point scale how closely they identify with 20 statements related to state anxiety. Outcome measure: state anxiety level (20-80).
Video Face Recording Phase 2 Sleep Deprivation | 3 minute recording every 3 hours starting Day 14 at 0930 until Day 16 1830.
  An application through the smartphone provided to the participant will be utilized to test if facial images captured with the phone camera could be used to assess the alertness level of subjects under sleep deprivation. Participants will be asked to remain still for 3 minutes as staff sets up the smartphone on a tripod in front of the subject and will use an application to record the video with the phone's rear camera. Staff will start the recording and the application will automatically stop the recording after 3 minutes. Will be used to test if facial images captured with phone camera could be used to assess alertness level of subjects under sleep deprivation
Video Face Recording Phase 3 Recovery | 3 minute recording every 3 hours on Day 17 at 0930, 1230, and 1530.
  An application through the smartphone provided to the participant will be utilized to test if facial images captured with the phone camera could be used to assess the alertness level of subjects under sleep deprivation. Participants will be asked to remain still for 3 minutes as staff sets up the smartphone on a tripod in front of the subject and will use an application to record the video with the phone's rear camera. Staff will start the recording and the application will automatically stop the recording after 3 minutes. Will be used to test if facial images captured with phone camera could be used to assess alertness level of subjects under sleep deprivation
Karolinska Sleepiness Scale (KSS) Phase 2 Sleep Deprivation | Task duration ~15 seconds, every 3 hours starting Day 14 at 0930 until Day 16 1830.
  To evaluate effects of sleep schedule on subjective sleepiness. Volunteers are presented with a 9-point sleepiness scale on a computer monitor (1=very alert, 3=alert, 5=neither alert nor sleepy, 7=sleepy (but not fighting sleep), 9=very sleepy (fighting sleep) and select the number on the scale that best reflects their current level of subjective sleepiness. Outcome measure: Number representing sleepiness (1-9)
Karolinska Sleepiness Scale (KSS) Phase 3 Recovery | Task duration ~15 seconds, every 3 hours on Day 17 at 0930, 1230, and 1530.
  To evaluate effects of sleep schedule on subjective sleepiness. Volunteers are presented with a 9-point sleepiness scale on a computer monitor (1=very alert, 3=alert, 5=neither alert nor sleepy, 7=sleepy (but not fighting sleep), 9=very sleepy (fighting sleep) and select the number on the scale that best reflects their current level of subjective sleepiness. Outcome measure: Number representing sleepiness (1-9)
Fatigue Visual Analog Scale (FVAS) Phase 2 Sleep Deprivation | Task duration ~15 seconds, every 3 hours starting Day 14 at 0930 until Day 16 1830.
  Measures fatigue on a continuous sliding scale from not fatigued to very fatigued. Subjects choose level of fatigue most closely corresponding to current level of fatigue. Outcome measure: fatigue level (0-100).
Fatigue Visual Analog Scale (FVAS) Phase 3 Recovery | Task duration ~15 seconds, every 3 hours on Day 17 at 0930, 1230, and 1530.
  Measures fatigue on a continuous sliding scale from not fatigued to very fatigued. Subjects choose level of fatigue most closely corresponding to current level of fatigue. Outcome measure: fatigue level (0-100).
Self-Assessment Manikin (SAM) Phase 2 Sleep Deprivation | Task duration: ~30 seconds every 3 hours starting Day 14 at 0930 until Day 16 1830.
  Measures levels of valence, arousal and dominance using a 7 point pictorial scale. Subjects are instructed to select which pictorial depiction most closely corresponds to current levels of valence, arousal, and dominance. Outcome measures: Valence, Arousal, and Dominance Levels (1-9)
Self-Assessment Manikin (SAM) Phase 3 Recovery | Task duration: ~30 seconds every 3 hours on Day 17 at 0930, 1230, and 1530.
  Measures levels of valence, arousal and dominance using a 7 point pictorial scale. Subjects are instructed to select which pictorial depiction most closely corresponds to current levels of valence, arousal, and dominance. Outcome measures: Valence, Arousal, and Dominance Levels (1-9)
Actigraphy | Throughout the entire study (~17.5 days)
  To determine amount and timing of sleep/wake periods during all phases of the study. Except for epochs that may be removed manually if they are determined to contain artifact, actigraphy records will be automatically scored by computer as either "sleep" or "wake" using the algorithms provided by the various manufacturers. Subjects will wear the actigraph continuously during Phases 1, 2, and 3. Outcome measures: Total sleep time, sleep latency, as well as raw epoch-by-epoch activity data, and heart rate (when available).

OTHER OUTCOMES:
Sleep period polysomnographic (PSG) measurements with video | During scheduled TIB periods (~2300 Day 13 to ~0700 Day 14 and ~2100 hrs on Day 16 to ~0900 hrs on Day 17) = ~20 hours of PSG recording per participant
  During in-laboratory periods while sleeping; PSG with video will be recorded continuously to assess and quantify sleep duration prior to the sleep deprivation period (Recording 1 - from ~2300 Day 13 to ~0700 Day 14) and to assess the effects of sleep loss on subsequent sleep architecture and document that recovery sleep was obtained prior to release from the study (Recording 2 - from ~2100 hrs on Day 16 to ~0900 hrs on Day 17). Outcome measures: total sleep time, sleep latency
Caffeine Use Tracking | ~30 seconds or less per entry as needed across Phase 1
  To monitor normal caffeine consumption during Phase 1. Subjects will track caffeine use using the app on the smartphone provided.These data will be utilized to individualize the 2B-Alert model for a participant.
Sleep Tracking | ~1 minute, once per day during Phase 1
  Monitor self-reported sleep duration during Phase 1. Subjects will log sleep duration using app on the smartphone provided. These data will be utilized to individualize the 2B-Alert model for a participant and compare against actigraphy data.
Beck Depression Inventory (BDI) | Administered at screening
  The BDI is a self-administered questionnaire with 21 questions. It provides a measure of a person's trait level of depression.
Horne-Ostberg Morningness-Eveningness (MEQ) | Administered at screening
  The MEQ is a 19-item questionnaire which assesses individual differences in the time of day a person prefers to carry out various activities, and classifies people as morning-type (M-type), neither-type (N-type) or evening-type (E-type) individuals.
Spielberger State-Trait Anxiety Inventory - Trait (STAI-T) | Administered at screening
  The STAI-T is a 20-item self-report questionnaire which assesses an individual's trait anxiety. The items are rated on a four-point scale. Higher scores indicate greater anxiety
NEO Five-Factor Inventory (NEO-FFI) | Administered at screening
  The NEO-FFI is a shortened version of the NEO PI-R, designed to give quick, reliable, and valid measures of the five domains of adult personality. The 60 items are rated on a five-point scale across five factors: Neuroticism, Extraversion, Openness to experience, Agreeableness, and Conscientiousness
Tridimensional Personality Questionnaire Harm Avoidance (TPQ-HA) | Administered at screening
  The Harm Avoidance scale of the TPQ is a 34-question true-false inventory to assess the stable personality trait of harm avoidance. Those volunteers with high harm avoidance scores are often more anxious and tense, avoid risk, and recover slowly from stress. Low harm avoidance score, on the other hand, indicate a volunteer is likely to engage in high risk behavior, be confident, and recover quickly from stress.
Connor-Davidson Resilience Scale (CD-RISC) | Administered at screening
  The CD-RISC comprises of 25 items, each rated on a 5-point scale (0-4), with higher scores reflecting greater resilience. The reliability, validity, and factor analytic structure of the scale have been evaluated, and reference scores for different study samples have been calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona, Tucson, Arizona, United States

REFERENCES:
- [Derived] Subramaniyan M, Vital-Lopez FG, Doty TJ, Anlap I, Killgore WDS, Reifman J. Personalized alertness prediction using video-based ocular and facial features. Sleep. 2025 Nov 10;48(11):zsaf149. doi: 10.1093/sleep/zsaf149. PMID 40457721